CLINICAL TRIAL: NCT06009796
Title: The Effects of Various Rapid Palatal Expansion Appliances on Dentoskeletal, Dentoalveolar, Nasal and Airway Resistance: A Prospective, Randomized Controlled Trial
Brief Title: The Effects of Various Rapid Palatal Expansion Appliances on Dentoskeletal, Dentoalveolar, Nasal and Airway Resistance
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: TC Erciyes University (Other)
Responsible Party: Principal Investigator, Ahmet Yağcı, PROFESSOR, TC Erciyes University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: TDH-2022-12101
Record Dates: First submitted 2023-08-16; First posted 2023-08-24 (Actual); Last update posted 2023-08-24 (Actual); Status verified 2023-08

CONDITIONS: Transverse Maxillary Deficiency
Keywords: Maxillary expansion; Respiratory polygraphy; Rhinomanometry; MARPE

STUDY DESIGN:
Intervention Model Description: Fifty eight patients were divided into 4 groups: FCRPE group (n: 15, 15.6 ± 1,1 years of age), MMRPE group (n:14, 15.3 ± 0,9 years of age), MARPE group (n:14, 15.7 ± 1,1 years of age), Control group (n:15, 15.4 ± 1,0 years of age). Polygraphy for respiratory evaluation, rhinomanometry for nasal airway resistance, study model and posteroanterior radiographs (PA) to measure dentoalveolar and dentoskeletal effects were used. Respiratory polygraphy, rhinomanometry, study model, and posteroanterior radiographs were obtained prior to treatment and after 3 months of expansion. Paired t tests and independent-sample t tests were used to compare the expansion appliances.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Full Coverage Rapid Palatal Expansion (FCRPE) group: (Active Comparator): Impressions were taken from the maxilla using alginate to obtain study models. In the obtained study model, a 10 mm hyrax expansion screw (Dentarum®, Germany) was placed at the midline as close to the palate as possible and parallel to the occlusal plane. The vestibular, occlusal, and palatal surfaces of all maxillary teeth are covered in acrylic, and this acrylic support extends toward the median palatal suture in the palatal region. Under pressure, the acrylic appliance was polymerized.
  Interventions: Device: Tooth Tissue Borne Rapid Palatal Expansion
- Modified McNamara Rapid Palatal Expansion (MMRPE) Group: (Active Comparator): Impressions were taken from the maxilla using alginate to obtain study models. In the obtained study model, a 10 mm hyrax expansion screw (Dentarum®, Germany) was placed at the midline as close to the palate as possible and parallel to the occlusal plane. The vestibular, occlusal, and palatal surfaces of the posterior maxillary teeth are covered in acrylic, and this acrylic support extends toward the median palatal suture in the palatal region. Under pressure, the acrylic appliance was polymerized.
  Interventions: Device: Tooth Tissue Borne Rapid Palatal Expansion
- Miniimplant Assisted Rapid Palatal Expansion (MARPE) Group (Active Comparator): The MARPE appliance was composed of a central expansion jackscrew (Dentarum), 4 tubes, 2 bands on the upper first molars to facilitate placement of the appliance, and 1.5-mm diameter stainless steel arms extending to the premolar teeth. Soldered stainless steel tubes (internal diameter: 2.0 mm; external diameter: 3.0 mm; length: 2.0 mm) served as guides for miniscrew placement. The size of the screws (PSM) was chosen as 1.8 mm in diameter and 11 mm in length, considering the 2 mm height of the tubes, 1 to 2 mm gap between the appliance and the palate surface, 1 to 2 mm gingiva thickness, and 5 to 6 mm length required for the bicortical placement of the screw in the bone.
  Interventions: Device: Tooth Bone Borne Rapid Palatal Expansion
- Control Group (No Intervention): A control group in the same age, without maxillary constriction was also added to our study.Polygraphy for respiratory evaluation, rhinomanometry for nasal airway resistance were used. Polygraphy and rhinomanometry measurements were obtained at the beginning of the follow-up and at the end of the 4-month follow-up period.

INTERVENTIONS:
Device: Tooth Tissue Borne Rapid Palatal Expansion — In all rapid palatal expansion groups, the appliances were cis bonded after being made by the same technician. The expansion screw was turned twice a day until the desired width was achieved.
  Arms: Full Coverage Rapid Palatal Expansion (FCRPE) group:; Modified McNamara Rapid Palatal Expansion (MMRPE) Group:
Device: Tooth Bone Borne Rapid Palatal Expansion — After the Marpe appliance was attached, 4 miniscrews were applied to the midline of the palate with a miniscrew driver. The expansion screw was turned twice a day until the desired width was achieved.
  Arms: Miniimplant Assisted Rapid Palatal Expansion (MARPE) Group

SUMMARY:
This study aims to evaluate the effects of dentoalveolar, dentoskeletal, nasal resistance, and airway changes by applying rapid palatal expansion appliances in patients with maxillary constriction and the post-pubertal growth spurt stage.

DETAILED DESCRIPTION:
Fifty eight patients were divided into 4 groups. The first group (n: 15, 15.6 ± 1,1 years of age) was Full Coverage Rapid Palatal Expansion (FCRPE). The second group ( n:14, 15.3 ± 0,9 years of age) was Modified McNamara Rapid Palatal Expansion (MMRPE). The third group (n:14, 15.7 ± 1,1 years of age) was Miniimplant Assisted Rapid Palatal Expansion (MARPE). The fourth group (n:15, 15.4 ± 1,0 years of age) was control group. Polygraphy for respiratory evaluation, rhinomanometry for nasal airway resistance, study model, and posteroanterior radiographs (PA) to measure dentoalveolar and dentoskeletal effects were used. Respiratory polygraphy, rhinomanometry, study model, and posteroanterior radiographs were obtained prior to treatment and after 3 months of expansion. Paired t tests and independent-sample t tests were used to compare the expansion appliances.

ELIGIBILITY:
Inclusion Criteria:

* With a unilateral or bilateral morphological lateral crossbite
* Whose first molars and premolars had completely erupted at pretreatment
* With maxillary constriction of more than 4 mm and less than 10 mm
* Who were going through the post-pubertal growth spurt stage based on hand-wrist radiographs
* Individuals with a body mass index of 18-24
* Individuals with an ANB angle between 0º and 4º

Exclusion Criteria:

* craniofacial anomalies
* compliance problems
* systemic or genetic disease
* previous orthodontic treatment history

Ages: 14 Years to 17 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 58 (Actual)
Dates: Start 2022-11-11 (Actual); Primary Completion 2023-03-14 (Actual); Study Completion 2023-07-12 (Actual)

PRIMARY OUTCOMES:
Rhinomanometry Measurement Parameters (Pa/cm3/sn ) | up to 1 year
  -Total Nasal Resistance(Pa/cm3/sn ): In our study, total nasal resistance was measured with a rhinomanometry device.
Polygraphy Measurement Parameters (event/hour) | up to 1 year
  - Apnea-Hypopnea Index (event/hour) : In our study, Apnea-Hypopnea Index(AHI) was measured with a polygraphy device. - Oxygen Desaturation index (De SPO2) : In our study, De SPO2 was measured with a polygraphy device.

SECONDARY OUTCOMES:
Postero-anterior Measurement Parameters(mm) | up to 1 year
  * NCB-NCB': Distance between right and left nasal cavity borders(mm)
  * JP-JP' : Distance between right and left jugal processes(mm)
  * AGP-AGP' : Distance between right and left antagonial points(mm)
Model Measurement Parameters(mm) | up to 1 year
  * C-C : Distance between cusp crests of canines(mm)
  * C'-C' : Distance between cingulum of canines(mm)
  * M1-M1 : The distance between buccal tubercles of first molar(mm)
  * M1'-M1' : The distance between the lingual tubercles of first molar(mm)

CONTACTS AND LOCATIONS:
Overall Officials: Ahmet YAGCI, PROFESSOR, Study Director — Erciyes University Faculty of Dentistry
Locations (1):
- Erciyes University Faculty of Dentistry ,Department of Orthodontics, Kayseri, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Lagravere MO, Major PW, Flores-Mir C. Skeletal and dental changes with fixed slow maxillary expansion treatment: a systematic review. J Am Dent Assoc. 2005 Feb;136(2):194-9. doi: 10.14219/jada.archive.2005.0141. PMID 15782523
- [Background] Lee KJ, Park YC, Park JY, Hwang WS. Miniscrew-assisted nonsurgical palatal expansion before orthognathic surgery for a patient with severe mandibular prognathism. Am J Orthod Dentofacial Orthop. 2010 Jun;137(6):830-9. doi: 10.1016/j.ajodo.2007.10.065. PMID 20685540
- [Background] Seeberger R, Kater W, Schulte-Geers M, Davids R, Freier K, Thiele O. Changes after surgically-assisted maxillary expansion (SARME) to the dentoalveolar, palatal and nasal structures by using tooth-borne distraction devices. Br J Oral Maxillofac Surg. 2011 Jul;49(5):381-5. doi: 10.1016/j.bjoms.2010.05.015. Epub 2010 Jun 17. PMID 21683264